CLINICAL TRIAL: NCT02190318
Title: The Effects of Losartan and Spironolactone on Residual Renal Function Preservation in Peritoneal Dialysis Patients
Brief Title: Residual Renal Function Preservation in Peritoneal Dialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Hong Liu, deputy director of nephrology department, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-RENAL-IIS-2013-029
Record Dates: First submitted 2014-07-12; First posted 2014-07-15 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Renal Disease
Keywords: peritoneal dialysis；; residual renal function；; RAAS
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Losartan; Spironolactone

ARMS (4):
- Losartan (Experimental): Losartan is taken orally 100mg/d
  Interventions: Drug: Losartan
- spirolactone (Experimental): spirolactone is taken orally 20mg/d
  Interventions: Drug: spirolactone
- losartan in combination with spirolactone (Experimental): Losartan is taken orally 100mg/d and spirolactone is taken orally 20mg/d
  Interventions: Drug: Losartan; Drug: spirolactone
- blank control (Sham Comparator): patients with antihypertensives besides ACEI/ARBs and spirolactone.
  Interventions: Other: blank control

INTERVENTIONS:
Drug: Losartan
  Arms: Losartan; losartan in combination with spirolactone
Drug: spirolactone
  Arms: losartan in combination with spirolactone; spirolactone
Other: blank control
  Arms: blank control

SUMMARY:
Aldosterone blockade is useful in preserving residual renal function in patients on PD.The long term efficacy of dual blockade of the RAAS is better than monotherapy.

DETAILED DESCRIPTION:
Residual renal function has been proven to contribute to improved survival and quality of life of dialysis patients. It is now recognized as an important factor in the prognosis of PD.The RAAS system is involved in the development of renal diseases. Angiotensin II and aldosterone are vital in this process. The beneficial effect of angiotensin-converting enzyme inhibitor or angiotensin receptor blocker on residual renal function has been demonstrated in peritoneal dialysis patients. Unfortunately, neither ACE inhibition nor angiotensin receptor blocker fully supprsses aldosterone production. Now much focus has been placed on aldosterone antagonist.

ELIGIBILITY:
Inclusion Criteria:

* Patients who having been on PD continuously for one month, urine volume>600 ml/d, residual renal function>2ml/min/1.73m2, blood pressure>120/70mmHg, serum potassium levels<5.5mmol/l, stable clinical condition.

Exclusion Criteria:

* Patients with infectious systemic disease, peritonitis during the preceding 1 month, who had taken ACEI/ARBs in the 3 preceding months, spirolactone in the 2 preceding weeks, intolerance to ACEI/ARBs, CHF, MI, malignant hypertension and stroke within the preceding 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
residual renal function of peritoneal dialysis patients | From date of randomization until the date of dropping out of the study or death from any cause, whichever came first, assessed up to 12 months.

SECONDARY OUTCOMES:
peritoneal membrane function | From date of randomization until the date of dropping out of the study or death from any cause, whichever came first, assessed up to 12 months.
  peritoneal membrane function is measured by peritoneal equilibration test to test the type of peritoneal transport. Briefly, a standard 4-hour dwell period was used (first exchange of the day), using a 2.5% glucose concentration 2-L volume exchange. The patient used their usual overnight dialysis regimen, and both the overnight and test drainage volumes were measured.The dialysate:plasma ratio of creatinine at the completion of the 4-hour dwell period (D/Pcreat) was used as the estimate of low-molecular-weight solute transport.

CONTACTS AND LOCATIONS:
Locations (1):
- Changsha, Hunan, China

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138